CLINICAL TRIAL: NCT03254134
Title: Comparative Effectiveness and Safety Between Warfarin and Dabigatran Using Real World Claims Data of Japanese Non-valvular Atrial Fibrillation Patients
Brief Title: Comparative Effectiveness and Safety Between Warfarin and Dabigatran
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0288
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin; Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial Fibrillation: patients with atrial fibrillation
  Interventions: Drug: Warfarin; Drug: Dabigatran

INTERVENTIONS:
Drug: Warfarin — patients treated with warfarin
Drug: Dabigatran — patients treated with Dabigatran
  Other Names: PRADAXA

SUMMARY:
This is a comparative effectiveness and safety study of clinical events among patients taking either dabigatran or warfarin. There is no formal hypothesis to be tested, but rather to provide the estimates on the incidence of stroke and systemic embolism (effectiveness) and bleeding events (safety) using 95% confidence interval for comparison between those non0-valvular atrial fibrillation patients taking dabigatran vs. warfarin using a large, nation-wide claims data in Japan.

DETAILED DESCRIPTION:
This is a comparative effectiveness and safety study of clinical events among patients taking either dabigatran or warfarin. There is no formal hypothesis to be tested, but rather to provide the estimates on the incidence of stroke and systemic embolism (effectiveness) and bleeding events (safety) using 95% confidence interval for comparison between those non-valvular atrial fibrillation patients taking dabigatran vs. warfarin using a large, nation-wide claims data in Japan.

ELIGIBILITY:
Inclusion Criteria:

* patients aged >18 year-old with confirmed diagnosis of Non-Valvular Atrial Fibrillation (NVAF) (ICD 10 code I48)
* having a first prescription (index date) of either dabigatran or warfarin between 14 March 2011 to 30 June 2016
* having no prescription of any Oral Anticoagulants (OACs) for 12 months prior to the index date (this period is defined as the baseline period)

Exclusion Criteria:

* patients having less than 12 months of enrolment prior to the index date
* being dialysis or kidney transplant recipients in baseline period
* having either atrial flutter, valvular atrial fibrillation (AF)
* mechanical valve placement, rheumatic AF
* and/or mitral valve prolapse/regurge/stenosis in baseline period
* having record of deep vein thrombosis or pulmonary embolism < 6 months before AF diagnosis in baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients with atrial fibrillation contained in the Medical Data Vision (MDVI) database which is a Japanese, nationwide claims data containing approximately 16 million patients cumulatively. The data cut is between March 2011 to June 2016, and the patients in the MDV database are those who have visited DPC hospitals (diagnostic procedure combination, a lump-sum payment system based on disease diagnosis to be treated similar to Medicare/Medicaid in the USA) hospitals which provide acute in-patient, as well as outpatient care.
Sampling Method: Non-Probability Sample
Enrollment: 22490 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A non-interventional study based on existing health insurance claims data. 5,146 and 13,115 patients were prescribed dabigatran and warfarin.
Pre-assignment Details: The Japanese patients diagnosed as Non-Valvular Atrial Fibrillation (NVAF) and newly treated with dabigatran and warfarin in the real world Japanese setting between April 2010 and June 2016 using the Medical Data Vision (MDV) database.
Groups:
- Dabigatran: Patients prescribed dabigatran as the first Oral Anticoagulants (OACs) with nonvalvular atrial fibrillation.
- Warfarin: Patients prescribed warfarin as the first Oral Anticoagulants (OACs) with nonvalvular atrial fibrillation.
Period: Overall Study
Arm/Group | Dabigatran | Warfarin
Started | 5745 | 16745
Completed | 5146 | 13115
Not Completed | 599 | 3630
Not completed — Not eligible patients | 599 | 3630

BASELINE CHARACTERISTICS:
Population: Eligible patients who were prescribed dabigatran and warfarin as the first OACs
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Warfarin | Total
Number analyzed (Participants) | 5146 | 13115 | 18261
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Eligible patients who were prescribed dabigatran and warfarin as the first OACs
  Years | 72 (10) | 78 (10) | 76 (10)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Eligible patients who were prescribed dabigatran and warfarin as the first OACs
  Participants
    Female | 1695 | 5294 | 6989
    Male | 3451 | 7821 | 11272
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Stroke and Systemic Embolism (SE)
Description: Incidence rate of stroke and systemic embolism (SE).
Time Frame: From the index date to end of treatment with > 14 day grace period, switch to another OAC, end of continuous enrolment, end of study period or death, outcome event of stroke and systemic embolism, ie., up to 6.5 years.
Population: Eligible patient who were prescribed dabigatran and warfarin as the first OACs and matched 1: 1 using the propensity score matching (PSM).
Measure: Number; unit: per patient-year
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 4606 | 4606
per patient-year | 2.898 | 3.563
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; There was no formal hypothesis testing; Test type: Superiority; Hazard Ratio (HR) = 0.720, 95% CI 2-sided [0.534 to 0.970]; The hazard ratio of stroke for the dabigatran group as compared to the warfarin group and its 95% CI were estimated from the propensity score matched group using a Cox regression model with treatment group as the dependent variable

2. Secondary Outcome: Incidence Rate of Major Bleeding
Description: Incidence rate of major bleeding defined by any bleeding event associated with hospitalization claims and/or transfusion claims.
Time Frame: From the index date to end of treatment with > 14 day grace period, switch to another OAC, end of continuous enrolment, end of study period or death, outcome event of major bleeding, ie., up to 6.5 years.
Population: as for outcome 1
Measure: Number; unit: per patient-year
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 4606 | 4606
per patient-year | 0.639 | 1.128
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; There was no formal hypothesis testing; Test type: Superiority; Hazard Ratio (HR) = 0.549, 95% CI 2-sided [0.303 to 0.994]; The hazard ratio of systemic embolism for the dabigatran group as compared to the warfarin group and its 95% CI were estimated from the propensity score matched group using a Cox regression model with treatment group as the dependent variable

ADVERSE EVENTS:
Description: This is a cohort study using based on existing data; therefore, it is not feasible to make a causality assessment at the individual case level.
Arm/Group | Dabigatran | Warfarin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03254134/Prot_SAP_000.pdf